CLINICAL TRIAL: NCT04662801
Title: A Behavioral Treatment With Sequenced Adjunctive Pharmacotherapy for Weight Regain After Bariatric Surgery: A Pilot Study
Brief Title: Weight Regain Treatment Post-Bariatric Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: American Psychological Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2000029491
Record Dates: First submitted 2020-12-09; First posted 2020-12-10 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-10

CONDITIONS: Obesity, Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Behavioral Weight Loss (Experimental)
  Interventions: Behavioral: Behavioral Weight Loss (BWL); Behavioral: Early Responder: BWL continued
- Behavioral Weight Loss + Medication (Experimental)
  Interventions: Behavioral: Behavioral Weight Loss (BWL); Combination Product: Early Non-responder: BWL continued with medication added

INTERVENTIONS:
Behavioral: Behavioral Weight Loss (BWL) — All participants will receive twelve weeks of BWL treatment.
Behavioral: Early Responder: BWL continued — Participants categorized as experiencing early weight loss at the end of the first month of treatment will continue with BWL for the remainder of treatment.
  Arms: Behavioral Weight Loss
Combination Product: Early Non-responder: BWL continued with medication added — Participants categorized as not experiencing early weight loss at the end of the first month of treatment will continue BWL plus a weight loss medication (Naltrexone Bupropion) for the remainder of treatment.
  Arms: Behavioral Weight Loss + Medication

SUMMARY:
This study will examine behavioral and pharmacologic (Naltrexone+Bupropion) treatments for weight regain after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Be in the age range ≥18 years of age and ≤70 years of age
* Have a BMI ≥30 (or BMI ≥27 with a medical comorbidity) and ≤50 kg/m2
* Have had laparoscopic Roux-en-Y gastric bypass or sleeve gastrectomy
* Experiencing weight regain after bariatric surgery
* Be an otherwise healthy subject without uncontrolled medical problems, as determined by the study physician and medical co-investigators (physical examination, laboratory studies).
* Read, comprehend, and write English at a sufficient level to complete study-related materials.
* Provide a signed and dated written informed consent prior to study participation.
* Be available for participation in the study for up to 3 months.

Exclusion Criteria:

* Has a predisposition to seizures (e.g., subject with a history or evidence of seizure disorder, febrile seizures during childhood, brain tumor, cerebrovascular disease, or significant head trauma; has a family history of idiopathic seizure disorder or is currently being treated with medications or treatment regimens that lower seizure threshold).
* Has a history of anorexia nervosa or history of bulimia nervosa.
* Is currently taking a medication that is a contraindication to NB medication (e.g., MAOI, opiates).
* Is currently using other medications for weight loss.
* Has a history of allergy or sensitivity to bupropion or naltrexone.
* Has a co-existing psychiatric condition that requires hospitalization or more intensive treatment (such as bipolar mood disorders, psychotic illnesses, or severe depression)
* Has untreated hypertension with a seated systolic blood pressure > 160 mmHg, diastolic blood pressure > 100 mmHg, or heart rate > 100 beats/minute.
* Has a history of congenital heart disease, cardiovascular disease, cardiac arrhythmias requiring medication, or a history of cerebrovascular pathology including stroke.
* Has current uncontrolled hypertension.
* Has current uncontrolled Type I or Type II diabetes mellitus.
* Has untreated hypothyroidism with a TSH > 1.5 times the upper limit of normal for the test laboratory with repeat value that also exceeds this limit.
* Has gallbladder disease.
* Has a history of severe renal, hepatic, neurological, chronic pulmonary disease, or any other unstable medical disorder.
* Has a recent history of drug or alcohol dependence (since having bariatric surgery).
* Is currently in active treatment for eating or weight loss.
* Is currently participating in another clinical study in which the subject is or will be exposed to an investigational or a non-investigational drug or device.
* Is breast-feeding or is pregnant or is not using a reliable form of birth control.
* Reports active suicidal or homicidal ideation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Behavioral Weight Loss | Behavioral Weight Loss + Medication
Started | 12 | 10
Completed | 9 | 7
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Weight Loss | Behavioral Weight Loss + Medication | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.17 (11.01) | 46.5 (7.71) | 49.05 (9.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 9 | 7 | 16
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Body Mass Index
Description: BMI is calculated using measured height and weight- kg/m2.
Time Frame: Post-treatment (3 months)
Population: Participants with complete data at follow up.
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Behavioral Weight Loss | Behavioral Weight Loss + Medication
Number analyzed (Participants) | 9 | 7
kg/m2 | 39.12 (4.57) | 40.48 (4.89)

2. Secondary Outcome: Eating Disorder Psychopathology
Description: Eating-disorder psychopathology is a continuous variable as assessed by the global score of the Eating Disorder Examination/Eating Disorder Examination-Questionnaire. Scores range from 0-6 (0=no eating-disorder psychopathology; 6=severe eating-disorder psychopathology).
Time Frame: Post-treatment (3 months)
Population: Participants with complete data at follow up- 1 participant did not complete questionnaires in the Behavioral Weight Loss + Medication group at follow up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Weight Loss | Behavioral Weight Loss + Medication
Number analyzed (Participants) | 9 | 6
units on a scale | 1.53 (0.80) | 1.46 (0.94)

3. Secondary Outcome: Food Craving
Description: Food craving will be assessed by the Food Craving Inventory (FCI). FCI scores range from 1-5, with higher scores indicative of greater craving.
Time Frame: Post-treatment (3 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Weight Loss | Behavioral Weight Loss + Medication
Number analyzed (Participants) | 9 | 6
units on a scale | 1.65 (0.49) | 1.57 (0.29)

4. Secondary Outcome: Depressive Symptoms
Description: Depressive symptoms will be assessed by the Patient Health Questionnaire-9. The range is 0-27, which higher scores indicative of greater depressive symptomatology
Time Frame: Post-treatment (3 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Weight Loss | Behavioral Weight Loss + Medication
Number analyzed (Participants) | 9 | 6
units on a scale | 3.89 (5.21) | 3.67 (2.58)

ADVERSE EVENTS:
Time Frame: Up to 3 months
Description: Adverse events were collected for both arms however, the on label listed potential side effects for the drug were used to assess participants in the '+ drug' arm systematically.
Arm/Group | Behavioral Weight Loss | Behavioral Weight Loss + Medication
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 0/12 | 7/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Behavioral Weight Loss (N=12) | Behavioral Weight Loss + Medication (N=10)
Diarrhea (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 0 | 4
Nausea (Gastrointestinal disorders) | 0 | 5
Dizziness (General disorders) | 0 | 3
Dry mouth (General disorders) | 0 | 5
Headache (General disorders) | 0 | 3
Insomnia (General disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/01/NCT04662801/Prot_SAP_000.pdf